CLINICAL TRIAL: NCT00815594
Title: Bleb Vascularity Change After Subconjunctival Injection of Bevacizumab
Brief Title: Bleb Vascularity Change After Subconjunctival Injection Bevacizumab
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Wang NingLi, Beiing Tongren hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008TR-LX-001
Record Dates: First submitted 2008-12-29; First posted 2008-12-30 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Bleb Vascularity; Conjunctival Scarring
Keywords: bleb; vascular change; bevacizumab; trabeculectomy; Bleb vascularity associated with increased scarring activity; Conjunctival scarring finally leads to the obstruction of the fistula tract created by the filtering surgery; the recombinant human anti-VEGF antibody could inhibit angiogenesis of conjunctiva.
MeSH Terms: conditions — Blister | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab — 0.05ml, 1.25mg

SUMMARY:
The occurrence of conjunctival scarring finally leads to the obstruction of the fistula tract created by the filtering surgery. Vascular endothelial growth factor is thought to be a key role in the formation of conjunctival scar, which play a pivotal role in the wound-healing process. So it seems that the recombinant human anti-VEGF antibody could inhibit angiogenesis, and reduce the conjunctival vascular formation in the wound-healing process after glaucoma filtering surgery.

ELIGIBILITY:
Inclusion Criteria:

* Glaucoma patients after trabeculectomy whose bleb is hyperaemia

Exclusion Criteria:

* Affected eye has normal IOP
* Not allergic with Avastin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-03 (Estimated); Study Completion 2009-05 (Estimated)

PRIMARY OUTCOMES:
bleb vascular change | one day, one week, one month

CONTACTS AND LOCATIONS:
Overall Officials: Liu Xuan, M.D., Principal Investigator — An ophthalmologist in Tongren hospital
Locations (1):
- Tongren hospital, Beijing, Beijing Municipality, China